CLINICAL TRIAL: NCT05317260
Title: Prognostic Relevance of Fatty Liver Disease for Patients With Chronic Hepatitis B
Brief Title: Steatohepatitis in Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Phunchai Charatcharoenwitthaya, Associated Professor, Mahidol University
Other Study IDs: 043/2560(EC2)
Record Dates: First submitted 2022-03-11; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Fatty Liver; Chronic Hepatitis b
MeSH Terms: conditions — Fatty Liver; Hepatitis B, Chronic | interventions — Antiviral Agents; Nucleosides

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — All liver biopsies were stained with Hematoxylin and Eosin, and Masson's trichrome. In cases of faded tissue slides, stored paraffin-embedded tissue block will be cut and re-stained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic hepatitis B patients without hepatic steatosis: Patients with chronic hepatitis B will be defined as the non-steatosis group if they had histological evidence of visible lipid droplets in hepatocytes less than 5%.
  Interventions: Drug: Antiviral Agents
- Chronic hepatitis B with steatosis but no steatohepatitis: Patients with chronic hepatitis B will be categorized as the steatosis but not steatohepatitis group if they had histological evidence of visible lipid droplets in hepatocytes more than 5% in the absence of steatohepatitis feature.
  Interventions: Drug: Antiviral Agents
- Chronic hepatitis B patients with steatohepatitis: Patients with chronic hepatitis B will be classified as the steatohepatitis group if they had histological evidence of steatosis, hepatocyte ballooning, mixed lobular acute and chronic inflammation, and intra-acinar perisinusoidal fibrosis according to Brunt's classification.
  Interventions: Drug: Antiviral Agents

INTERVENTIONS:
Drug: Antiviral Agents — The type of antiviral agents for the individual patient was selected by physicians based on a policy to reimburse a patient's health and comorbidity.
  Other Names: Nucleoside analogue; Nucleotide analogue; Peginterferon

SUMMARY:
Fatty liver disease is increasingly recognized in patients with chronic hepatitis B (CHB). Whether concurrent fatty liver disease affects the long-term outcomes of CHB is unclear. The investigators performed a longitudinal study to investigate the prognostic relevance of concurrent fatty liver disease for patients with CHB receiving antiviral therapy.

DETAILED DESCRIPTION:
Chronic hepatitis B virus (HBV) infection is a global public health problem affecting more than 250 million people at high risk of death from cirrhosis and liver cancer. The goal of therapy for patients with chronic hepatitis B (CHB) is to improve survival and quality of life by preventing disease progression to cirrhosis, hepatic decompensation, and hepatocellular carcinoma (HCC). This can be achieved by elimination of HBV or sustained suppression of viral replication with antiviral treatment. In recent years, accompanied by the growing prevalence of obesity, fatty liver disease is commonly observed in patients with CHB. The prevalence of the fatty liver disease is approximately 14-67% in Asian individuals with CHB, similar to Western countries. The coexistence of CHB and hepatic steatosis, particularly steatohepatitis, can aggravate liver damage and increase the risk of fibrosis. A recent histological study showed a significant association between steatohepatitis and advanced fibrosis in CHB patients.

Fatty liver disease has been shown to increase the risk of fibrosis progression in patients with CHB receiving antiviral treatment. According to a follow-up study of cirrhotic patients treated with tenofovir disoproxil fumarate for CHB, patients with possible concurrent NAFLD were less likely to have fibrosis regression despite viral suppression. Likewise, another prospective study showed that lower body mass index was independently associated with fibrosis regression in CHB patients who achieved undetectable HBV viral load during long-term nucleoside analogue therapy. Hence, monitoring the development of unfavorable outcomes is recommended in this population. However, there are limited data on the impact of concurrent fatty liver disease on clinical outcomes (e.g., cirrhotic complications, HCC, and death) during comprehensive treatment for CHB. Therefore, this longitudinal cohort study aimed to determine the effect of concurrent fatty liver disease on overall survival and liver-related complications among CHB patients receiving antiviral therapy to improve our understanding of the prognostic value of concurrent fatty liver disease in these patients.

METHODS The investigators conduct a retrospective analysis of a prospectively collected database of patients with chronic HBV infection who underwent a liver biopsy between 2002 and 2008 at the Faculty of Medicine Siriraj Hospital in Bangkok, Thailand. This cohort includes only patients who had at least moderate necroinflammation and/or liver fibrosis stage 2 or higher according to the METAVIR system and have been treated with antiviral agents. Patients will be excluded from analysis if they had co-infection with hepatitis C virus or human immunodeficiency virus; had the presence of alcohol dependence; had follow-up data less than six months in our clinic; had no available liver histology for review; had intermittent or persistent HBV DNA >2000 IU/ml after stopping antiviral agents during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All CHB patients who had significant histologic features, defined as at least moderate necroinflammation and/or liver fibrosis stage 2 or higher according to the METAVIR system, required antiviral therapy and have been managed in our institution.
* HBV-treated patients who had achieved undetectable HBV DNA or hepatitis B surface antigen (HBsAg) loss during antiviral therapy, and those who had hepatitis B e antigen (HBeAg) seroconversion with serum HBV DNA persistently <2,000 IU/ml and normalization of aminotransferase levels after discontinuing antiviral therapy.

Exclusion Criteria:

* Patients who had viremia >2000 IU/ml after stopping antiviral agents will be excluded.
* Patients with a history of alcohol dependence or co-infections with hepatitis C virus or human immunodeficiency virus before liver biopsy will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis B patients who underwent liver biopsy during 2002-2008 and then received antiviral therapy. The studied patients had achieved undetectable HBV DNA or hepatitis B surface antigen (HBsAg) loss during antiviral therapy, and those who had hepatitis B e antigen (HBeAg) seroconversion with serum HBV DNA persistently <2,000 IU/ml and normalization of aminotransferase levels after discontinuing antiviral therapy. According to Brunt's classification, patients will be categorized into three groups, including non-steatosis, steatosis but no steatohepatitis, and steatohepatitis groups based on the histological features of the liver specimens.
Sampling Method: Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Overall mortality | From date of liver biopsy until the date of liver transplantation or date of death from any cause, whichever came first, assessed up to 22 years
  Death from any cause

SECONDARY OUTCOMES:
Liver-related complications | From date of liver biopsy until the date of first documented liver-related complications, whichever came first, assessed up to 22 years
  Liver-related complications such as hepatocellular carcinoma, spontaneous bacterial peritonitis, variceal hemorrhage, portosystemic encephalopathy, and hepatorenal syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Phunchai Charatcharoenwitthaya, MD., Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analyzed during the current study are not publicly available due to our University's institutional review boards (IRB) and the health insurance portability and accountability act (HIPAA) privacy rule but are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Schweitzer A, Horn J, Mikolajczyk RT, Krause G, Ott JJ. Estimations of worldwide prevalence of chronic hepatitis B virus infection: a systematic review of data published between 1965 and 2013. Lancet. 2015 Oct 17;386(10003):1546-55. doi: 10.1016/S0140-6736(15)61412-X. Epub 2015 Jul 28. PMID 26231459
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. No abstract available. PMID 29405329
- [Background] Sarin SK, Kumar M, Lau GK, Abbas Z, Chan HL, Chen CJ, Chen DS, Chen HL, Chen PJ, Chien RN, Dokmeci AK, Gane E, Hou JL, Jafri W, Jia J, Kim JH, Lai CL, Lee HC, Lim SG, Liu CJ, Locarnini S, Al Mahtab M, Mohamed R, Omata M, Park J, Piratvisuth T, Sharma BC, Sollano J, Wang FS, Wei L, Yuen MF, Zheng SS, Kao JH. Asian-Pacific clinical practice guidelines on the management of hepatitis B: a 2015 update. Hepatol Int. 2016 Jan;10(1):1-98. doi: 10.1007/s12072-015-9675-4. Epub 2015 Nov 13. PMID 26563120
- [Background] Powell EE, Wong VW, Rinella M. Non-alcoholic fatty liver disease. Lancet. 2021 Jun 5;397(10290):2212-2224. doi: 10.1016/S0140-6736(20)32511-3. Epub 2021 Apr 21. PMID 33894145
- [Background] Eslam M, Sanyal AJ, George J; International Consensus Panel. MAFLD: A Consensus-Driven Proposed Nomenclature for Metabolic Associated Fatty Liver Disease. Gastroenterology. 2020 May;158(7):1999-2014.e1. doi: 10.1053/j.gastro.2019.11.312. Epub 2020 Feb 8. PMID 32044314
- [Background] Charatcharoenwitthaya P, Pongpaibul A, Kaosombatwattana U, Bhanthumkomol P, Bandidniyamanon W, Pausawasdi N, Tanwandee T. The prevalence of steatohepatitis in chronic hepatitis B patients and its impact on disease severity and treatment response. Liver Int. 2017 Apr;37(4):542-551. doi: 10.1111/liv.13271. Epub 2016 Oct 31. PMID 27740738
- [Background] Mak LY, Seto WK, Hui RW, Fung J, Wong DK, Lai CL, Yuen MF. Fibrosis evolution in chronic hepatitis B e antigen-negative patients across a 10-year interval. J Viral Hepat. 2019 Jul;26(7):818-827. doi: 10.1111/jvh.13095. Epub 2019 Apr 16. PMID 30895682
- [Background] Marcellin P, Gane E, Buti M, Afdhal N, Sievert W, Jacobson IM, Washington MK, Germanidis G, Flaherty JF, Aguilar Schall R, Bornstein JD, Kitrinos KM, Subramanian GM, McHutchison JG, Heathcote EJ. Regression of cirrhosis during treatment with tenofovir disoproxil fumarate for chronic hepatitis B: a 5-year open-label follow-up study. Lancet. 2013 Feb 9;381(9865):468-75. doi: 10.1016/S0140-6736(12)61425-1. Epub 2012 Dec 10. PMID 23234725
- [Background] Seto WK, Fung J, Cheung KS, Mak LY, Hui RW, Liu KS, Lai CL, Yuen MF. Body-mass index is associated with fibrosis regression during long-term nucleoside analogue therapy in chronic hepatitis B. Aliment Pharmacol Ther. 2016 Nov;44(10):1071-1079. doi: 10.1111/apt.13804. Epub 2016 Sep 22. PMID 27659292
- [Background] Kleiner DE, Brunt EM, Van Natta M, Behling C, Contos MJ, Cummings OW, Ferrell LD, Liu YC, Torbenson MS, Unalp-Arida A, Yeh M, McCullough AJ, Sanyal AJ; Nonalcoholic Steatohepatitis Clinical Research Network. Design and validation of a histological scoring system for nonalcoholic fatty liver disease. Hepatology. 2005 Jun;41(6):1313-21. doi: 10.1002/hep.20701. PMID 15915461
- [Background] Brunt EM, Janney CG, Di Bisceglie AM, Neuschwander-Tetri BA, Bacon BR. Nonalcoholic steatohepatitis: a proposal for grading and staging the histological lesions. Am J Gastroenterol. 1999 Sep;94(9):2467-74. doi: 10.1111/j.1572-0241.1999.01377.x. PMID 10484010

DOCUMENTS (2):
  • Study Protocol (2021-12-31): https://cdn.clinicaltrials.gov/large-docs/60/NCT05317260/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-31): https://cdn.clinicaltrials.gov/large-docs/60/NCT05317260/SAP_001.pdf